CLINICAL TRIAL: NCT03433729
Title: A Randomized Controlled Trial to Assess the Impact of an Agenda Setting Form in a Respiratory Outpatient Clinic: Are Patients More Likely to Perceive That Their Important Issues Are Discussed and Does the Form Improve Clinic Efficiency?
Brief Title: Patient Agenda Setting and Clinic Efficiency in Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Jonathan Fuld, Consultant Physician, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A092512
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Respiratory Tract Diseases
Keywords: Outpatient Clinics, Hospital; Humans; Outcome Assessment (Health Care); Patient Outcome Assessment; Patient satisfaction; Hospitalists; Secondary care
MeSH Terms: conditions — Respiratory Tract Diseases; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Agenda Form (Experimental): Patient Agenda form: Patients receive an agenda form to use before their consultation.
  Interventions: Other: Patient agenda form
- Usual care (No Intervention): Patients' appointment continues as usual.

INTERVENTIONS:
Other: Patient agenda form — On arrival at the clinic patients are given an agenda form to prompt them to think about what issues they wished to discuss with their doctor. The form contains a prompt list of items they can tick, free space to write their own items, and a prompt to consider what is the most important issue for them and what they would like to happen before they leave their clinic appointment.
  Arms: Patient Agenda Form

SUMMARY:
The purpose of the study is to determine whether patients who use a prompt sheet to identify their important issues before they see a doctor are more likely to feel that their important issues have been discussed during their consultation. The study will be conducted in a respiratory outpatient clinic.

DETAILED DESCRIPTION:
Evidence suggests that most patients come to a consultation with issues they wish to raise, but they may not actually raise them and clinicians may not elicit them. This can adversely affect the consultation outcome, e.g. through misunderstandings, unwanted prescriptions, non-adherence and unnecessary follow-ups. In a review of methods used before consultations to help patients address their information needs Kinnersely et al. (2009) found that there were small but statistically significant increases in patient satisfaction and the number of questions patients asked, and no effect on consultation length. However, they identified several gaps in the evidence including the need to assess a wider range of outcome measures, to identify the impact of the methods on the types of questions asked and the need to measure consultation length accurately.

This study aims to assess the impact of a written agenda form in a respiratory outpatient clinic. The form prompts the patient to identify their questions and issues, provides a list of frequently asked questions and invites the patient to write down the issues they wish to discuss with their doctor. We wish to identify whether use of the form increases the extent to which patients perceive that their important issues are discussed in the consultation. We will also assess whether patients feel more able to raise these issues and get the outcome they wanted, their confidence to manage their condition and consultation length.

The study is a randomised controlled trial (RCT) with a sample size of 158 patients. On arrival at the clinic patients will be randomly allocated to either the intervention group (who will receive an agenda form) or to standard practice. Patient reported outcomes will be collected after the patient has seen the doctor and consultation times will be recorded by an independent observer outside the consultation room.

ELIGIBILITY:
Inclusion Criteria:

* have an outpatient appointment at one of the designated clinics
* are able to understand the Patient Information Sheet and complete the agenda form and the feedback form, or are accompanied by a person who meets this criteria and who is willing to complete the form on the patient's behalf
* willing and able to give informed consent for participation in the study

Exclusion Criteria:

* No further criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who, on leaving their outpatient appointment, strongly agree with the statement "My doctor discussed the issues that were important to me" where options are strongly agree, agree, disagree, strongly disagree. | Immediately after consultation with the doctor

SECONDARY OUTCOMES:
The proportion of patients who strongly agree with the statement "I got the outcome I wanted from my consultation" where options are strongly agree, agree, disagree, strongly disagree. | Immediately after consultation with the doctor
The proportion of patients who strongly agree with the statement "I felt able to raise issues that were important to me with my doctor" where options are strongly agree, agree, disagree, strongly disagree | Immediately after consultation with the doctor
Patient confidence to manage their condition following the consultation, rated on a scale of 0-10 where 0 equals no confidence and 10 equals maximum confidence | Immediately after consultation with the doctor
Length of consultation | Immediately after consultation with the doctor

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Fuld, MD ChB, PhD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom